CLINICAL TRIAL: NCT03448731
Title: Phase II Clinical Trial of Doxycycline 50 mg or 100 mg Daily for the Prevention of Skin Toxicity in Patients With Metastatic Colorectal Cancer Treated With Anti-EGFR and Chemotherapy
Brief Title: Skin Toxicity in Patients With Metastatic Colorectal Cancer Treated With Anti-EGFR and Chemotherapy (DERMIA)
Acronym: DERMIA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fundacion CRIS de Investigación para Vencer el Cáncer (Other)
Collaborators: Amgen (Industry); Apices Soluciones S.L. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DERMIA; 2017-004413-98 (EudraCT Number)
Record Dates: First submitted 2018-02-19; First posted 2018-02-28 (Actual); Last update posted 2020-04-08 (Actual); Status verified 2020-04

CONDITIONS: Skin Toxicity
MeSH Terms: interventions — Doxycycline; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Doxycycline (Experimental): Doxycycline 50 mg p.o. daily during 6 weeks
  Interventions: Drug: Doxycycline 50Mg Tablet

INTERVENTIONS:
Drug: Doxycycline 50Mg Tablet — Doxycycline administered p.o once daily at a 50 mg dose for 6 weeks beginning on Day -1

SUMMARY:
Clinical evidence has suggested that sub-antimicrobial doses of doxycycline may have the potential to treat inflammatory lesions of acne. The efficacy of doses below 100 mg/day of doxycycline in the prevention of skin toxicity in patients with treated with Epidermal Growth Factor Receptor (EGFR)-targeted therapies has never been studied. Therefore, the aim of the present study is to describe the efficacy of doxycycline 50 or 100 mg per day in the prevention of skin toxicity in patients with metastatic Colorectal cancer (mCRC) treated with anti-EGFR in combination with chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman at least 18 years old
* Capable of understanding, signing and dating an informed consent approved by an Independent Ethics Committee (IEC)
* Histologically confirmed adenocarcinoma of the colon or rectum in patients with initially unresectable metastatic (M1) disease
* Wild-type RAS tumour status confirmed before study inclusion at local institution
* Patients who have a treatment plan based on FOLFOX + anti-EGFR or FOLFIRI + anti-EGFR, as first-line treatment of mCRC
* Eastern Cooperative Oncology Group (ECOG) performance status ≤2
* Adequate bone marrow function: neutrophils ≥1.5 x109/L; platelets ≥100 x109/L; haemoglobin ≥9 g/dL
* Hepatic, renal and metabolic function as follows: Total bilirubin count ≤1.5 x upper limit of normal (ULN), Alanine aminotransferase (ALT) and Aspartate aminotransferase (AST) <5 x ULN; Renal function, calculated as creatinine clearance or 24-hour creatinine clearance ≥50 mL/min; Magnesium > lower limit of normal (LLN)

Exclusion Criteria:

* History of prior or concurrent central nervous system (CNS) metastases
* History of another primary cancer, except: curatively treated in situ cervical cancer, or curatively resected non-melanoma skin cancer, or other primary solid tumour curatively treated with no known active disease present and no treatment administered for ≥5 years before treatment initiation
* Known hypersensitivity to tetracyclines
* Prior chemotherapy or other systemic anticancer therapy for treatment of metastatic colorectal carcinoma
* Prior adjuvant chemotherapy for colorectal cancer terminated less than 6 months before metastatic disease was diagnosed
* Unresolved toxicities of a previous systemic treatment that, in the opinion of the investigator, cause the patient unfit for inclusion
* Prior anti-epidermal growth factor receptor (EGFR) antibody therapy (e.g., cetuximab), antivascular endothelial growth factor (VEGF) or treatment with small molecule EGFR inhibitors (e.g., erlotinib)
* Prior hormonal therapy, immunotherapy or approved or experimental antibody/proteins ≤30 days before inclusion.
* Significant cardiovascular disease including unstable angina or myocardial infarction within 12 months before initiating study treatment or a history of ventricular arrhythmia
* History of interstitial pneumonitis or pulmonary fibrosis or evidence of interstitial pneumonitis or pulmonary fibrosis on baseline chest computed tomography (CT)
* Treatment for systemic infection within 14 days before the start of study treatment
* Acute or subacute intestinal occlusion and/or active inflammatory bowel disease or other bowel disease that causes chronic diarrhoea (defined as grade ≥ 2 diarrhoea according to Common Terminology Criteria for Adverse Events (CTCAE)
* Clinically significant peripheral sensory neuropathy
* Evidence of previous acute hypersensitivity reaction, of any grade, to any component of the treatment
* History of Gilbert disease or known dihydropyrimidine deficiency syndrome
* Recent gastroduodenal ulcer to be active or uncontrolled
* Recent pulmonary embolism, deep vein thrombosis, or other significant venous event
* Pre-existing bleeding diathesis and/or coagulopathy with exception of well-controlled anticoagulation therapy
* Recent major surgical procedure, open biopsy, or significant traumatic injury not yet recovered from prior major surgery
* History of any disease that may increase the risks associated with study participation or may interfere with the interpretation of study results.
* Known positive test for human immunodeficiency virus infection, hepatitis C virus, chronic active hepatitis B infection
* Any disorder that compromises the patient's ability to provide written informed consent and/or comply with study procedures
* Any investigational agent within 30 days prior to inclusion
* Pregnant or breastfeeding woman
* Surgery (excluding diagnostic biopsy or placement of a central venous catheter) and/or radiotherapy within 28 days prior to inclusion in the study.
* Male or female of childbearing age who do not agree with taking adequate contraceptive precautions, i.e. use contraception double barrier (e.g. diaphragm plus condoms) or abstinence during the course of the study and for 6 months after the last administration of study drug for women and 1 month for men
* The patient is unwilling or unable to meet the requirements of the study. Psychological, geographical, familial or sociological conditions that potentially prevent compliance with the study protocol and follow-up schedule. These conditions should be discussed with the patient before inclusion in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2018-05-10 (Actual); Primary Completion 2020-04-06 (Actual); Study Completion 2020-04-06 (Actual)

PRIMARY OUTCOMES:
Efficacy in the prevention of skin toxicity | During 6-week skin treatment
  Monitoring of skin toxicities graded according to National Cancer Institute Common Terminology Criteria for Adverse Events

SECONDARY OUTCOMES:
Quality of life of patients during the treatment | Up to 7 weeks
  Change in Dermatology Life Quality Index (DLQI) score
Incidence of Treatment-Emergent Adverse Events | Up to 6 weeks
  Number of adverse events per patient

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Ramirez-Daffós, MD, Principal Investigator — Hospital Universitario Puerta del Mar
Locations (8):
- Spain (8):
  - Hospital Punta Europa, Algeciras
  - Hospital Puerta del Mar, Cadiz
  - Hospital Puerto Real, Cadiz
  - Hospital San Pedro de Alcántara, Cáceres
  - Hospital Clinico San Cecilio, Granada
  - Hospital Juan Ramón Jiménez, Huelva
  - Hospital de Jerez, Jerez de la Frontera
  - Hospital Virgen Macarena, Seville

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ramirez-Daffos P, Jimenez-Orozco E, Bolanos M, Gonzalez Astorga B, Rubiales S, Ceballos-Barbancho E, Rodriguez Garcia JM, Reina JJ. A phase 2 study for evaluating doxycycline 50 mg once daily and 100 mg once daily as preemptive treatment for skin toxicity in patients with metastatic colorectal cancer treated with an anti-EGFR and chemotherapy. Support Care Cancer. 2022 Oct;30(10):8081-8088. doi: 10.1007/s00520-022-07254-5. Epub 2022 Jul 1. PMID 35776185